CLINICAL TRIAL: NCT05082155
Title: Continuous Erector Spinae Plane Blocks to Treat Postoperative Pain After Open Gynecologic Procedures Via a Low Transverse (Pfannenstiel) Incision: A Randomized, Triple-masked, Placebo-controlled, Split-body Clinical Trial
Brief Title: Continuous Erector Spinae Plane Blocks to Treat Postoperative Pain After Open Gynecologic Procedures Via a Low Transverse (Pfannenstiel) Incision
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: surgeons stopped doing procedures
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bilateral cESPB for GYN Surg
Record Dates: First submitted 2021-10-02; First posted 2021-10-18 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Surgical Incision; Pain, Postoperative; Pain, Acute
MeSH Terms: conditions — Surgical Wound; Pain, Postoperative; Acute Pain | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a split-body study in which each study subject receives both treatments: one on each side of the body. Which treatment is applied to which side of the body is randomized (and masked).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will be created by the University of California San Diego Investigational Drug Service. Investigational pharmacists will prepare all study solutions as determined by the randomization list. Bupivacaine and normal saline are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff will be masked to treatment group assignment for the duration of the enrollment and data collection period. Unmasking will not occur until statistical analysis is complete (termed "triple masking").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Right sided catheter bupivacaine 0.25% and left sided catheter normal saline (Experimental): This is a split body study. Bilateral erector spinae plane catheters will be inserted and study fluid is administered bilaterally. Bupivacaine 0.25 will be administered through the right-sided catheter while normal saline will be administered through the left-sided catheter. Both infusion pumps will be programmed to deliver a basal infusion of 1 mL/h and an automatic intermittent bolus of 20 mL every 4 hours.
  Interventions: Drug: Bupivacaine 0.25%; Drug: Normal Saline
- Right sided catheter normal saline and left sided catheter bupivacaine 0.25% (Experimental): This is a split body study. Bilateral erector spinae plane catheters will be inserted and study fluid is administered bilaterally. Normal saline will be administered through the right-sided catheter while bupivacaine 0.25% will be administered through the left-sided catheter. Both infusion pumps will be programmed to deliver a basal infusion of 1 mL/h and an automatic intermittent bolus of 20 mL every 4 hours.
  Interventions: Drug: Bupivacaine 0.25%; Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine 0.25% — Bupivacaine 0.25% will be delivered as a basal infusion of 1 mL/h and an automatic intermittent bolus of 20 mL every 4 hours.
Drug: Normal Saline — Normal saline will be delivered as a basal infusion of 1 mL/h and an automatic intermittent bolus of 20 mL every 4 hours.
  Other Names: Placebo

SUMMARY:
Open gynecologic surgery can be very painful. With the goal of minimizing the use of opioids (with undesired side effects and potential for abuse), the investigators often administer a type of peripheral nerve block in which the investigators put local anesthetic-or, numbing medicine-near the nerves that go to the surgical area which helps to numb the area and decrease pain following surgery. These blocks with a single-injection of local anesthetic are called erector spinae plane (ESP) blocks, and they are applied on each side of the body since each injection affects only that one side. However, the numbing medication typically lasts for only 16-20 hours. For other peripheral nerve blocks, this duration can be increased with the insertion of a catheter-a tiny tube smaller than a piece of spaghetti-followed by an infusion of additional local anesthetic. However, the effects of the various peripheral nerve blocks are determined by the anatomy and physiology of the specific peripheral nerve, with an infusion resulting in dramatic benefits for one nerve yet having no effect for another. The potential benefits and risks of adding a catheter and subsequent local anesthetic infusion to a single-injection ESP block remain unknown. The investigatorstherefore propose a randomized, triple-masked, placebo-controlled, split-body clinical trial to determine the potential benefits and risks of adding the infusion to single-injection ESP blocks.

DETAILED DESCRIPTION:
Open gynecologic surgery can be significantly painful. With the goal of minimizing the use of opioids (with undesired side effects and potential for abuse), the investigators frequently administer bilateral single-injection erector spinae plane (ESP) blocks which help to numb the surgical area and decrease postoperative pain. However, the numbing medication typically lasts for only 8-18 hours. For other peripheral nerve blocks, this duration can be increased with the insertion of a percutaneous catheter-a tiny tube smaller than a piece of spaghetti-followed by an infusion of additional local anesthetic. However, the effects of the various peripheral nerve blocks are determined by the anatomy and physiology of the specific peripheral nerve, with an infusion resulting in dramatic benefits for one nerve yet having no effect for another. The potential benefits and risks of adding a catheter and subsequent local anesthetic infusion to a single-injection ESP block remain unknown.

The investigators therefore propose a randomized, triple-masked, placebo-controlled, split-body clinical trial to determine the potential benefits and risks of adding the infusion to single-injection ESP blocks. Patients undergoing gynecologic surgery via a low transverse (Pfannenstiel) incision who already have bilateral ESP blocks as part of their analgesic plan will be offered enrollment. Participants will have bilateral catheters inserted through the same block needles used for their single-injections, followed by perineural administration of bupivacaine on one side and normal saline on the other (determined randomly and in a triple-masked fashion).

This will be a single-center, randomized, triple-masked, placebo-controlled, split-body human subjects clinical trial.

Enrollment. Participants will be consenting adults undergoing open gynecologic surgery via a low transverse incision. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current Institutional Review Board-approved informed consent form. The study population of interest includes women of all races and socioeconomic status. Inclusion and exclusion criteria are listed in section #10 below. Of note, the investigators will be using local anesthetic, perineural catheters, and infusion pumps as approved/cleared by the Food and Drug Administration and do not plan to research a possible change of indication or use of these medications/devices as part of this research project.

Preoperative Procedures. Following written, informed consent, the investigators will record baseline anthropometric information (age, sex, height, and weight) that is already provided by all patients having surgery. Participants will have a peripheral intravenous catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned sitting. Intravenous midazolam and fentanyl will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area of insertion will be sterily prepared and a clear, sterile, fenestrated drape applied. In the sitting position and with ultrasound guidance, after subcutaneous local infiltration with lidocaine- a 17g Tuohy and 5-10 ml of saline with 1:200,000 epinephrine will be used to identify the correct plane, as defined by a hyperechoic shadow of the 10th transverse process and erector spine muscle immediately superficial. Once appropriate needle tip location is confirmed, a perineural catheter will be inserted under ultrasound guidance. This procedure will be repeated on the contralateral side.

Following negative aspiration, 20 mL of 0.25% bupivacaine with 1:200,000 of epinephrine will be injected via both catheters with sonographic confirmation of local anesthetic spread. Blocks will be considered successful if, within 30 minutes, the participant experiences decreased sensation to cold temperature over the level of the ipsilateral 10th thoracic dermatome at the level of anterior axillary line. Failed blocks/catheters will be successfully replaced or the participant withdrawn from the study.

Treatment Group Assignment. The right-sided catheter will be randomized to one of two treatment groups: bupivacaine 0.25% or normal saline ("study infusate"). The contralateral side will receive the other possible study infusate (either bupivacaine 0.25% or normal saline). Therefore, each participant will receive both treatments-one on each side-and act as their own control.

Randomization will be stratified for benign vs. malignant surgical indication, in block sizes of 4. The randomization list will be created by the University of California San Diego Investigational Drug Service. Investigational pharmacists will prepare all study solutions as determined by the randomization list. Bupivacaine and normal saline are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff will be masked to treatment group assignment for the duration of the enrollment and data collection period. Unmasking will not occur until statistical analysis is complete (termed "triple masking").

Study intervention. Perineural study infusate administration will be initiated within the operating or recovery rooms. Both infusion pumps will be programmed to deliver a basal infusion of 1 mL/h and an automatic intermittent bolus of 20 mL every 4 hours. This dose of bupivacaine is well-within the standard maximum dose at our institution for perineural local anesthetic administration for other truncal locations such as the paravertebral space. No patient-controlled bolus dose will be included. For any cases of inadvertent premature catheter dislodgement, the subject may opt to have the catheter replaced.

Perineural catheters will be removed by healthcare providers upon study infusate reservoir exhaustion (approximately 50 hours) or just prior to hospital discharge-whichever comes first.

Postoperative analgesics. In addition to the perineural study infusate, subjects will receive standard-of-care oral and intravenous postoperative analgesics which can include acetaminophen, ibuprofen, gabapentin, and opioids (this is surgeon- and patient-dependent). Therefore, all patients of this study-regardless of the treatment arm they are randomized to-will continue to receive current usual and customary analgesia: all will receive the same combination of acetaminophen, ibuprofen, gabapentin, opioids, and a single-injection erector spinae plane block as they would regardless of study participation.

Outcome measurements (end points). The investigators have selected outcome measures that have established reliability and validity, with minimal inter-rater discordance, and are recommended for pain-related clinical trials by the World Health Organization and the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus statement. All data collection will be through standard UCSD nursing/therapy EPIC notes and patient interviews in-person during hospitalization or via a telephone call. All pain scores will be recorded for each side of the body (trunk) at each time point, measured using the Numeric Rating Scale.

The overall objective of the proposed research is to determine the risks and benefits of adding a continuous erector spinae plane (ESP) block to a single-injection ESP in patients undergoing open gynecologic surgery via a low transverse incision.

Specific Aim 1: To determine the risks and benefits of adding a continuous ESP block to a single-injection ESP the day following open gynecologic surgery.

Hypothesis 1.1: Analgesia will be improved the day following surgery with the addition of a continuous ESP block as measured with the Numeric Rating Scale ("average" pain included in the Brief Pain Inventory pain domain) [primary end point].

Hypothesis 1.2: Breakthrough pain will be decreased the day following surgery with the addition of a continuous ESP block as measured with the Numeric Rating Scale ("worst" pain included in the Brief Pain Inventory pain domain).

Hypothesis 1.3: Pain during coughing will be decreased the day following surgery with the addition of a continuous ESP block as measured with the Numeric Rating Scale.

Specific Aim 2: To determine the risks and benefits on postoperative day 2 of adding a continuous ESP block to a single-injection ESP following open gynecologic surgery.

Hypothesis 2.1: Analgesia will be improved on postoperative day 2 with the addition of a continuous ESP block as measured with the Numeric Rating Scale ("average" pain included in the Brief Pain Inventory pain domain).

Hypothesis 2.2: Breakthrough pain will be decreased on postoperative day 2 with the addition of a continuous ESP block as measured with the Numeric Rating Scale ("worst" pain included in the Brief Pain Inventory pain domain).

Hypothesis 2.3: Pain during coughing will be decreased on postoperative day 2 with the addition of a continuous ESP block as measured with the Numeric Rating Scale.

Analysis Approach Baseline characteristics by randomized side (bupivacaine to the left vs bupivacaine to the right) will be summarized with means, standard deviations, and quartiles. Balance between groups will be assessed. Specifically, standardized differences will be calculated using Cohen's d whereby the difference in means or proportions is divided by the pooled standard deviation estimates. Any key variables (age, sex, height, weight, and BMI) with an absolute standardized difference >0.78 (with 1.96×√(2/12.5)=0.78 [with a sample size of 25, the investigators expect about 12.5 randomized to left vs right]) will be noted and included in a linear regression model to obtain an estimate of the treatment effect adjusted for the imbalanced covariate(s). If residuals from the linear regression indicate violations of key assumptions (i.e. homoscedasticity or Gaussian distribution), data transformations and/or alternative generalized linear models will be applied as appropriate. If no imbalance is detected, the primary analysis will proceed by a one-sample Wilcoxon test applied to the difference between paired observations (bupivacaine minus saline). Secondary outcomes will also be analyzed by one-sample Wilcoxon test, or linear models (or generalized linear models) as appropriate to adjust for any imbalanced covariates.

The primary analysis will exclude patients from the analysis if their low transverse incision is unexpectedly converted to a vertical incision following randomization. The investigators will compare the characteristics of these excluded participants compared to the primary analysis population, and also report results for the full intention-to-treat population (all randomized participants).

Gatekeeping strategy Hypotheses will be tested with strong control of the familywise error rate at 5%.

Testing begins with a single primary hypotheses H11. If this test is significant at the 0.05 level, that alpha is passed on to other hypotheses. For example, if the p-value for H12 is less than 0.025, but the p-value for H13 is not, then H13 can be tested at the 0.025 + 0.025/2 = 0.0375 level. If both H12 and H13 are rejected, no alpha is spent, and the investigators go on to similarly test H21, H22, and H23. If a given test does not reach local significance, alpha is spent and cannot be passed along to hypotheses.

Simulated Power for NRS Power is estimated by simulations assuming a minimum clinically meaningful effect: NRS difference scores (bupivacaine minus saline, with negative scores favoring bupivacaine) are distributed with a median of -1 and interquartile range (IQR) -3 to 0. This IQR for a bilateral difference is consistent with unilateral IQRs (6 to 6 and 7 to 7) reported in Boules et al. (2020). A sample size of n=25 individuals would provide 84% power to detect such an effect with two-sided α=0.05.

Along with cancelled surgeries and drop-out cases, the investigators anticipate requiring the consenting of 35 subjects to produce a data set consisting of a minimum of 25 subjects to be included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing open gynecologic surgery via a low transverse incision;
2. Analgesic plan includes bilateral single-injection ESP blocks; and
3. Age 18 years or older.

Exclusion Criteria:

1. Morbid obesity as defined by a body mass index > 40 (BMI=weight in kg / [height in meters]2);
2. Renal insufficiency (abnormal preoperative creatinine or eGFR );
3. Chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks);
4. History of opioid abuse;
5. Any comorbidity which results in moderate or severe functional limitation;
6. Inability to communicate with the investigators or hospital staff;
7. Pregnancy;
8. Planned intrathecal opioids;
9. Incarceration;
10. Known allergy to any study medication; and
11. Any contraindication to perineural catheter insertion (e.g., infection at the catheter insertion site).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
"Average" pain during postoperative day 1 as measured using the numeric rating scale, collected postoperative day 1 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale | Postoperative day 1 (00:01 through afternoon data-collection time point)
  The "average" pain measured using the numeric rating scale, collected postoperative day 1 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain

SECONDARY OUTCOMES:
Maximum pain during postoperative day 1 which is the highest pain measured using the numeric rating scale, collected postoperative day 1 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0=no pain, 10=worst pain | Postoperative day 1 (00:01 through afternoon data-collection time point)
  The highest pain measured using the numeric rating scale, collected postoperative day 1 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
Pain during coughing, postoperative day 1 which is the highest pain experienced during coughing using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0= no pain and 10= worst pain | Postoperative Day 1 at the time of the data collection time point
  The highest pain experienced during coughing using the numeric rating scale, collected postoperative day 1. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
"Average" pain during postoperative day 2 which is the "average" pain measured using the numeric rating scale, collected postoperative day 2 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10=worst pain | Postoperative day 2 (00:01 through afternoon data-collection time point)
  The "average" pain measured using the numeric rating scale, collected postoperative day 2 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst pain
Maximum pain during postoperative day 2 which is the highest pain experienced during coughing using the numeric rating scale, collected postoperative day 2. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain | Postoperative day 2 (00:01 through afternoon data-collection time point)
  The highest pain experienced during coughing using the numeric rating scale, collected postoperative day 2. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
Pain during coughing, postoperative day 2 which is tthe highest pain experienced during coughing using the numeric rating scale, collected postoperative day 2. pain | Postoperative Day 2 at the time of the data collection time point
  The highest pain experienced during coughing using the numeric rating scale, collected postoperative day 2. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
"Average" pain during postoperative day 3 which is the "average" pain measured using the numeric rating scale, collected postoperative day 3 for the time since midnight. It is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst pain | Postoperative day 3 (00:01 through afternoon data-collection time point)
  The "average" pain measured using the numeric rating scale, collected the postoperative day 3 for the time since midnight. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
Maximum pain during postoperative day 3 which is the highest pain experienced during coughing using the numeric rating scale, collected postoperative day 3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain | Postoperative day 3 (00:01 through afternoon data-collection time point)
  The highest pain experienced during coughing using the numeric rating scale, collected postoperative day 3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
Pain during coughing, postoperative day 3 which is the highest pain experienced during coughing using the numeric rating scale, collected postoperative day 3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst pain | Postoperative Day 3 at the time of the data collection phone call
  The highest pain experienced during coughing using the numeric rating scale, collected postoperative day 3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
"Current" pain during postoperative days 1-3 which is the current pain experienced using the numeric rating scale, collected postoperative days 1-3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain | Postoperative Days 1-3 at the time of the data collection time point
  The current pain experienced using the numeric rating scale, collected postoperative days 1-3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
Least pain during postoperative days 1-3 which is the lowest pain experienced since midnight using the numeric rating scale, collected postoperative days 1-3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst pain | Postoperative day1 1-3 (00:01 through afternoon data-collection time point)
  The lowest pain experienced since midnight using the numeric rating scale, collected postoperative days 1-3. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain

OTHER OUTCOMES:
Surgical start time | Day of surgery
  Time of day recorded using military time
Surgical duration | Day of surgery
  The duration from surgical start until stop measured in hours and minutes
Indication for surgery | Day of surgery
  Reason the patient underwent the surgical procedure [e.g., benign vs. malignant tumor]
Opioid consumption | Postoperative Days 0-3
  Amount of opioids consumed daily and cumulatively measured in morphine equivalents
Infusion duration | Postoperative Days 0-3
  The time from the end of surgery until the catheters were removed
Hospital length of stay | Postoperative Days 0-3
  The day of discharge
Antiemetic use | Recovery room, postoperative days 0-2
  Any antiemetic medication consumed
Time to oral intake | Postoperative Days 0-3
  Day and time of first oral intake
Time to flatus | Postoperative Days 0-3
  Day and time of first postoperative flatus
Time to first bowel movement | Postoperative Days 0-3
  Day and time of first bowel movement
Subjective weakness of hip flexion and/or knee extension | Postoperative Days 1-3
  If (yes or no) patient feels like the muscles that flex the hip and/or extend the knee joints are weak
Number of participants with an intraoperative conversion to a vertical incision: study enrollment will be offered only to participants who are having a low, horizontal surgical incision; however, in rare cases the surgeons convert to a vertical incision | Day of surgery
  If the surgeon made a vertical incision intraoperatively
Number of participants with an inadvertent catheter dislodgment | Postoperative Days 0-3
  A catheter that was found dislodged from its original level at the skin

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD,MS, Principal Investigator — UCSD Medical Center
Locations (1):
- University Of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No